CLINICAL TRIAL: NCT04625959
Title: Optimizing Mindfulness and Acceptance Based Behavioral Treatment for Bulimia Nervosa and Binge Eating Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2001007570
Record Dates: First submitted 2020-09-16; First posted 2020-11-12 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Bulimia Nervosa; Bulimia; Atypical; Binge-Eating Disorder; Binge-Eating and Purging Type Anorexia Nervosa; Binge Eating
Keywords: Mindfulness and Acceptance Based Behavioral Treatments; Eating Disorders; Bulimia Nervosa; Binge Eating Disorder; Anorexia Nervosa Binge/Purge Type; Binge Eating
MeSH Terms: conditions — Bulimia Nervosa; Bulimia; Binge-Eating Disorder; Feeding and Eating Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: MOST: multiphase optimization strategy
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Base BT (Active Comparator): 16 weekly sessions of behavioral therapy.
  Interventions: Behavioral: Behavioral Therapy for Eating Disorders
- Base BT + Distress Tolerance (Experimental): 16 weekly sessions of behavioral therapy with distress tolerance components of MABTs.
  Interventions: Behavioral: MABT: Distress Tolerance
- Base BT + Emotion Regulation (Experimental): 16 weekly sessions of behavioral therapy with emotion regulation components of MABTs.
  Interventions: Behavioral: MABT: Emotion Modulation
- Base BT + Mindful Awareness (Experimental): 16 weekly sessions of behavioral therapy with mindful awareness components of MABTs.
  Interventions: Behavioral: MABT: Mindful Awareness
- Base BT + Values (Experimental): 16 weekly sessions of behavioral therapy with values components of MABTs.
  Interventions: Behavioral: MABT: Values
- Base BT + Distress Tolerance and Emotion Modulation (Experimental): 16 weekly sessions of behavioral therapy with emotion regulation and distress tolerance components of MABTs.
  Interventions: Behavioral: MABT: Emotion Modulation; Behavioral: MABT: Distress Tolerance
- Base BT + Distress Tolerance and Mindful Awareness (Experimental): 16 weekly sessions of behavioral therapy with distress tolerance and mindful awareness components of MABTs.
  Interventions: Behavioral: MABT: Mindful Awareness; Behavioral: MABT: Distress Tolerance
- Base BT + Distress Tolerance and Values (Experimental): 16 weekly sessions of behavioral therapy with distress tolerance and values components of MABTs.
  Interventions: Behavioral: MABT: Values; Behavioral: MABT: Distress Tolerance
- Base BT + Emotion Modulation and Mindful Awareness (Experimental): 16 weekly sessions of behavioral therapy with emotion regulation and mindful awareness components of MABTs.
  Interventions: Behavioral: MABT: Mindful Awareness; Behavioral: MABT: Emotion Modulation
- Base BT + Mindful Awareness and Values (Experimental): 16 weekly sessions of behavioral therapy with values and mindful awareness components of MABTs.
  Interventions: Behavioral: MABT: Mindful Awareness; Behavioral: MABT: Values
- Base BT + Emotion Modulation and Values (Experimental): 16 weekly sessions of behavioral therapy with emotion regulation and values components of MABTs.
  Interventions: Behavioral: MABT: Values; Behavioral: MABT: Emotion Modulation
- Base BT + EM, DT, MA (Experimental): 16 weekly sessions of behavioral therapy with emotion regulation, mindful awareness, and distress tolerance components of MABTs.
  Interventions: Behavioral: MABT: Mindful Awareness; Behavioral: MABT: Emotion Modulation; Behavioral: MABT: Distress Tolerance
- Base BT + DT, ER, and V (Experimental): 16 weekly sessions of behavioral therapy with emotion regulation, distress tolerance, and values components of MABTs.
  Interventions: Behavioral: MABT: Values; Behavioral: MABT: Emotion Modulation; Behavioral: MABT: Distress Tolerance
- Base BT + DT, MA, and V (Experimental): 16 weekly sessions of behavioral therapy with distress tolerance, mindful awareness, and values components of MABTs.
  Interventions: Behavioral: MABT: Mindful Awareness; Behavioral: MABT: Values; Behavioral: MABT: Distress Tolerance
- Base BT + ER, MA, and V (Experimental): 16 weekly sessions of behavioral therapy with emotion regulation, mindful awareness, and values components of MABTs.
  Interventions: Behavioral: MABT: Mindful Awareness; Behavioral: MABT: Values; Behavioral: MABT: Emotion Modulation
- Base BT + ER, MA, V, DT (Experimental): 16 weekly sessions of behavioral therapy with emotion regulation, mindful awareness, distress tolerance, and values components of MABTs.
  Interventions: Behavioral: MABT: Mindful Awareness; Behavioral: MABT: Values; Behavioral: MABT: Emotion Modulation; Behavioral: MABT: Distress Tolerance

INTERVENTIONS:
Behavioral: Behavioral Therapy for Eating Disorders — Change behaviors that maintain binge eating (e.g. rigid dietary restriction outside of binge episodes, irregular or chaotic eating patterns).
  Arms: Base BT
Behavioral: MABT: Mindful Awareness — Integrates behavioral treatment for eating disorders with a set of psychological strategies, specifically mindful awareness, designed to enhance self-regulation. Mindful awareness strategies include developing inner and outer wisdom, formal meditation, and shifting awareness to the present moment. Mindful awareness skills also include increasing awareness of thoughts, feelings, physical sensations, and hunger and fullness cues.
  Arms: Base BT + DT, MA, and V; Base BT + Distress Tolerance and Mindful Awareness; Base BT + EM, DT, MA; Base BT + ER, MA, V, DT; Base BT + ER, MA, and V; Base BT + Emotion Modulation and Mindful Awareness; Base BT + Mindful Awareness; Base BT + Mindful Awareness and Values
Behavioral: MABT: Values — Integrates behavioral treatment for eating disorders with a set of psychological strategies, specifically values, designed to enhance self-regulation. Values skills include identifying and clarifying values, living a values life, making values-consistent decisions, addressing competing values, values awareness, and using values to address negative moods.
  Arms: Base BT + DT, ER, and V; Base BT + DT, MA, and V; Base BT + Distress Tolerance and Values; Base BT + ER, MA, V, DT; Base BT + ER, MA, and V; Base BT + Emotion Modulation and Values; Base BT + Mindful Awareness and Values; Base BT + Values
Behavioral: MABT: Emotion Modulation — Integrates behavioral treatment for eating disorders with a set of psychological strategies, specifically emotion modulation, designed to enhance self-regulation. Emotion modulation skills include long-term habits for emotion regulation, coping strategies, crisis management, and cognitive reappraisal.
  Arms: Base BT + DT, ER, and V; Base BT + Distress Tolerance and Emotion Modulation; Base BT + EM, DT, MA; Base BT + ER, MA, V, DT; Base BT + ER, MA, and V; Base BT + Emotion Modulation and Mindful Awareness; Base BT + Emotion Modulation and Values; Base BT + Emotion Regulation
Behavioral: MABT: Distress Tolerance — Integrates behavioral treatment for eating disorders with a set of psychological strategies, specifically distress tolerance, designed to enhance self-regulation. Distress tolerance skills include psychological acceptance, uncoupling, willingness, and dealing with dirty distress.
  Arms: Base BT + DT, ER, and V; Base BT + DT, MA, and V; Base BT + Distress Tolerance; Base BT + Distress Tolerance and Emotion Modulation; Base BT + Distress Tolerance and Mindful Awareness; Base BT + Distress Tolerance and Values; Base BT + EM, DT, MA; Base BT + ER, MA, V, DT

SUMMARY:
The current study will use a full factorial design to identify the independent and combined effects of four core MABT components when combined with standard behavioral treatment for BN and BED. The primary aim of the study will be to evaluate the independent efficacy of Mindful Awareness, Distress Tolerance, Emotion Modulation, and Values-Based Decision Making on eating pathology (at posttreatment and at 6 and 12-month follow-ups). Secondary aims will be (1) to test target engagement of each MABT component, i.e., to confirm that each treatment component impacts both the variable which it targets and self-regulation and that improvements in these are associated with improvements in outcomes and (2) to test the hypotheses that the efficacy of each component is moderated by related baseline deficits in self-regulation (e.g. individuals with worse distress tolerance at baseline are most likely to benefit from conditions that include the Distress Tolerance component). A final exploratory aim will be to quantify the component interaction effects, which may be partially additive (because components overlap and/or there is diminishing return), fully additive, or synergistic (in that components may partially depend on each other).

ELIGIBILITY:
Inclusion Criteria:

1. Have experienced 12 or more loss of control episodes within the previous 3 months
2. Have a BMI above 16
3. Are located in the US and wiling/able to participate in remote treatment and assessments
4. Are able to give consent

Exclusion Criteria:

1. Are unable to fluently speak, write and read English
2. Have a BMI below 16
3. Are receiving treatment for an eating disorder
4. Require immediate treatment for medical complications as a result of eating disorder symptoms
5. Have a mental handicap, or are experiencing other severe psychopathology that would limit the participants' ability to comply with the demands of the current study (e.g. severe depression with suicidal intent, active psychotic disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Binge eating frequency assessed by the Eating Disorder Examination | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and 6-month and 1 year post-treatment follow-up assessment
  Frequency (number of days and number of instances) of binge eating over the past 28 days assessed by the Eating Disorder Examination
Eating Disorder Examination | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and 6 month and 1 year post-treatment follow-up assessment
  The Eating Disorder Examination is a semi-structured interview that measures eating pathology. The EDE yields four subscale scores: Restraint, Eating Concern, Shape Concern, and Weight Concern. The possible score range for each subscale is 0 to 6. The total score may also be reported (determined by averaging the subscale scores); the score range for the total score is also 0 to 6. For subscale scores and total score, higher scores indicate more severe pathology. The restraint sub-scale of the EDE will be used to assess utilization of skills related to reducing dietary restraint.
Remission Status | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and 6 month and 1 year post-treatment follow-up assessment
  Presence or absence of eating disorder diagnosis. Not in remission; in partial remission; or in full remission.

SECONDARY OUTCOMES:
Compensatory behavior frequency assessed by the Eating Disorder Examination (EDE) | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and 6 month and 1 year post-treatment follow-up assessment
  Frequency (number of days and number of instances) of compensatory behaviors assessed by the Eating Disorder Examination
BMI | Changes from each assessment time point throughout treatment (3 assessments over 16 weeks) and 6 month and 1 year post-treatment follow-up assessment
  kilogram/(meters^2), this is an outcome measure for participants with anorexia nervosa, binge/purge type

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Stratton Hall, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: For more information, send an email to EDresearch@drexel.edu or call (215) 553-7130 — http://drexel.edu/coas/academics/departments-centers/well-center/research/current-research-projects/